CLINICAL TRIAL: NCT07052929
Title: A Phase 1/2, Multicenter, Open-label, Dose Escalation and Expansion Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of ASP2957 in Male Participants With Invasive Ventilator-dependent X-linked Myotubular Myopathy
Brief Title: Study of ASP2957 in Male Participants With X-linked Myotubular Myopathy Who Need Ventilators
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2957-CL-0101; 2025-523213-29 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: X-Linked Myotubular Myopathy
Keywords: XLMTM; Recombinant Adeno-Associated Virus
MeSH Terms: conditions — Myopathies, Structural, Congenital | interventions — Methylprednisolone; Prednisolone; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 : ASP2957 Dose Escalation (Experimental): Participants will receive sequential dose levels of a single infusion of ASP2957 and immunosuppression prophylaxis including methylprednisolone, prednisolone and sirolimus.
  Interventions: Genetic: ASP2957; Drug: Methylprednisolone; Drug: Prednisolone; Drug: Sirolimus
- Part 2: ASP2957 Dose Expansion (Experimental): Participants will receive a single infusion of ASP2957 (dose selected in Part 1) and immunosuppression prophylaxis including methylprednisolone, prednisolone and sirolimus.
  Interventions: Genetic: ASP2957; Drug: Methylprednisolone; Drug: Prednisolone; Drug: Sirolimus

INTERVENTIONS:
Genetic: ASP2957 — Intravenous infusion
  Other Names: MyoAAV3.8 engineered capsid - myosin heavy chain kinase 7 - human myotubularin (MyoAAV3.8-MHCK7-hMTM1)
Drug: Methylprednisolone — Intravenous infusion
Drug: Prednisolone — Route of administration based on locally sourced product
Drug: Sirolimus — Route of administration based on locally sourced product

SUMMARY:
X-linked myotubular myopathy (XLMTM) is a rare and serious condition present at birth where the muscles do not work properly. There are currently no approved therapies for XLMTM.

The protein myotubularin is needed for muscle development, movement and breathing. A gene called MTM1 tells the body to make myotubularin. XLMTM is caused by changes, or mutations, in the MTM1 gene. Changes in the MTM1 gene cause low or no levels of myotubularin to be made, so the muscles do not work properly.

Gene therapy is a way of getting a healthy copy of a gene into the body. This allows the body's cells to make a normal protein that may reduce disease symptoms. Researchers have developed ASP2957 to get a healthy MTM1 gene into the body. This could help improve muscle development and function in young children with XLMTM.

In this study, ASP2957 will be given to humans for the first time.

ASP2957 has the healthy MTM1 gene inside a type of empty (killed) virus. The virus delivers the healthy MTM1 gene directly into cells in the body. It's possible that some boys may have antibodies to the virus if they have previously been infected with a similar virus. The antibodies could stop ASP2957 from working properly and cause an immune reaction to ASP2957. To prevent this, the boys will also be given medicines to lower the immune system.

The main aims of this study are to check the safety of ASP2957, how well it is tolerated, and to find a suitable dose of ASP2957.

The study was designed in 2 phases. In Phase 1, different small groups of boys will receive lower to higher doses of ASP2957. Each boy will receive a single infusion of ASP2957. Any medical problems will be recorded for each dose. This is done to find a suitable dose of ASP2957 to use in Phase 2.

In Phase 2, another small group of young boys will receive a single infusion of ASP2957. The most suitable dose of ASP2957 worked out from Phase 1 will be used.

The boys will be checked for up to 1 year after their single infusion of ASP2957. After this, there will be the option for the boys to join another study so they will continue to be checked longer term.

ELIGIBILITY:
Inclusion Criteria:

* Participant is projected to be ≤ 36 months of age at dosing.
* Participant has molecular genetic report from a CAP-approved testing facility at screening that confirms a diagnosis of XLMTM and harbors a "pathogenic" or "likely pathogenic" variant in the MTM1 gene as classified using the American College of Medical Genetics (ACMG) standards and guidelines for interpretation of sequence variants. Although samples will be sent to the sponsor central laboratory during screening for exploratory testing, results of this testing are not required for enrollment.
* Participant is ventilator-dependent and meets the following criteria:

  * Required respiratory support at birth
  * Requires ≥ 20 hours per day of invasive ventilator support (confirmed during screening)
  * Has a tracheostomy tube
* Participant has no evidence of hepatic peliosis, increased echogenicity or any other clinically important abnormal finding on liver ultrasound.
* Participant can receive immunosuppression per protocol.
* Participant's hepatobiliary laboratory measurements must meet the criteria during screening and for the 2-month retrospective assessment of participant's medical history:
* Participant's hematological laboratory measurements must meet the criteria during screening:
* Participant's parent(s) or legally authorized representative LAR(s) must provide documentation of being current with recommended immunization schedule according to regional guidelines.

  * If any immunization has not been administered, the medical reasons must be documented by the investigator along with medical risk associated with ASP2957 and immunosuppression administration. The sponsor will review the risk assessment with the investigator and determine the participant's eligibility for the study.
  * Immunizations requiring administration after inclusion in the study must be administered in accordance with regional guidelines for live, live attenuated and inactivated immunization prior to, during and after stopping immunosuppression with methylprednisolone, prednisolone and sirolimus. For an example of guidelines, see Centers for Disease Control and Prevention (CDC) General Best Practices Guidelines for Immunization.
  * Immunization of household contacts can be considered based on regional standards of care of individuals receiving immunosuppression regimens.
* Participant and participant's parent(s) or LAR(s) are willing and able to comply with study visits and study procedures.
* Participant's parent(s) or LAR(s) agree that the participant will not participate in another interventional study from the time of signing the Informed Consent Form (ICF) through week 52.
* Participant's parent(s) or LAR(s) is willing to transition the participant to a separate long-term follow-up study after study completion.

Exclusion Criteria:

* Participant born < 35 weeks gestation is still not term as per corrected age.
* Participant is nutritionally unstable with weight less than fifth percentile for age or has a vitamin A, E or K deficiency.
* Participant requires supplemental oxygen on a routine or chronic basis.

  * Note: The use of supplemental oxygen for acute, self-limited illnesses (for example, during hospitalization for pneumonia) shall not be exclusionary, provided the participant is neither acutely ill nor using supplemental oxygen at the time of screening.
* Participant currently has a clinically important respiratory infection or other clinically important active infection of any kind.
* Participant has an active viral or bacterial infection including, but not limited to, positive testing for:

  * tuberculosis (TB) using the QuantiFERON-TB test
  * Active hepatitis A virus (HAV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
  * Prior HBV or HCV virus infection due to the risk of reactivation associated with immunosuppression
  * human immunodeficiency virus type 1 (HIV-1) and human immunodeficiency virus type 2 (HIV-2)
  * coronavirus disease 2019 (COVID-19)
  * cytomegalovirus (CMV), including either positive CMV immunoglobulin G (IgG) or presence of detectable CMV DNA by quantitative polymerase chain reaction (PCR) at screening.
* Participant has any history of cholestatic liver dysfunction and/or treatment for cholestasis. If the participant is taking prophylactic treatment for cholestasis (e.g., ursodiol, cholestyramine, rifampin or other therapies) which has not been prescribed for cholestatic liver dysfunction, treatment must be discontinued for at least 4 weeks prior to signing the ICF.

  * Neonatal hyperbilirubinemia resolving within 4 weeks of birth in a full-term infant is not an exclusion.
* Participant has prior history of abnormal transaminases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST)) and/or abnormal bilirubin metabolism associated with ascites, jaundice (aside from neonatal hyperbilirubinemia) or gastrointestinal bleeding.
* Participant has a significant medical condition or life-threatening disease other than XLMTM that would interfere with adhering to protocol requirements or would increase the risk of immunosuppression and/or recombinant adeno-associated virus (rAAV) administration.
* Participant has musculoskeletal complications such as severe contractures and/or scoliosis that would limit the ability to observe improvements in neuromuscular function.

  * In participants with scoliosis, the Cobb angle must be < 40 degrees for study eligibility.
* Other than as required per protocol, participant has received or plans to receive systemic immunomodulating agents within 90 days before day 1 (use of inhaled corticosteroids to manage chronic respiratory conditions is allowed).
* Participant has previously received monoclonal antibodies of any type.

  * Exception: Monoclonal antibodies to prevent RSV are permitted, except for during the 4 weeks prior to the initiation of immunosuppression.
* Participant plans to have surgery within 12 weeks prior to day 1 through week 52 that may confound safety and efficacy data interpretation of the study intervention.

  * Exception: Standard of care surgical interventions such as gastrostomy, jejunostomy and Nissen fundoplication procedures are allowed.
* Participant received any treatment for cholestasis (e.g., ursodiol, cholestyramine, rifampin or other therapies) prior to signing the ICF.
* Participant is participating in another interventional study or has received an adeno-associated virus (AAV)-based gene therapy.
* Participant tests positive for anti-MyoAAV3.8 TAb, as determined by central laboratory testing.

  * Since very young children may have passive antibodies transferred in utero from the mother, participants ≤ 6 months of age who initially test positive for anti-MyoAAV3.8 total antibody (TAb) may be rescreened for study eligibility.
* Participant has a known or suspected contraindication or hypersensitivity to methylprednisolone, prednisolone, sirolimus or any components of the ASP2957 formulation.
* Participant has a contraindication to general anesthesia, magnetic resonance imaging (MRI) or muscle biopsy procedures.
* Any other reason that would render the participant unsuitable for participation in the study, including risk of non-adherence to the study assessments and protocol.

Max Age: 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | Up to week 52
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures. A TEAE is defined as an AE observed after administration of ASP2957.
Number of participants with adverse events of special interest (AESIs) | Up to week 52
  AESIs include myocardial-associated events, muscle abnormalities, hepatobiliary disorders, thrombocytopenia, TMA and life-threatening infections.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 52 weeks
  Number of participants with potentially clinically significant laboratory values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 52 weeks
  Number of participants with potentially clinically significant ECGs.
Number of participants with echocardiogram (ECHO) abnormalities and/or AEs | Up to 52 weeks
  Number of participants with potentially clinically significant ECHOs.
Number of participants with muscle magnetic resonance imaging (MRI) abnormalities and/or AEs | Up to 52 weeks
  Number of participants with potentially clinically significant muscle MRIs.
Number of participants with histopathology abnormalities and/or AEs from muscle biopsy | Up to 52 weeks
  Number of participants with potentially clinically significant histopathology from muscle biopsy.
Number of participants with physical examinations abnormalities and/or AEs | Up to 52 weeks
  Number of participants with potentially clinically significant physical examinations.

SECONDARY OUTCOMES:
Change from baseline in hours per day of ventilation support at week 52 | Baseline and up to week 52
  The hours of ventilation support will be collected.
ASP2957 vector deoxyribonucleic acid (DNA) in serum through week 52 | Up to week 52
  ASP2957 vector DNA will be recorded from serum samples collected.
ASP2957 vector DNA in muscle biopsy at week 52 | Week 52
  ASP2957 vector DNA will be recorded from muscle biopsy collected.
ASP2957 vector DNA in saliva | Up to week 52
  ASP2957 vector DNA will be recorded from saliva samples collected.
ASP2957 vector DNA in urine | Up to week 52
  ASP2957 vector DNA will be recorded from urine samples collected.
ASP2957 vector DNA in stool | Up to week 52
  ASP2957 vector DNA will be recorded from stool samples collected.
Anti-MyoAAV3.8 total antibody (TAb) | Up to week 52
  Anti-MyoAAV3.8 TAb will be recorded from serum samples collected
Anti-MyoAAV3.8 neutralizing antibody (NAb) | Up to week 52
  Anti-MyoAAV3.8 NAb will be recorded from serum samples collected.
Anti-myotubularin TAb | Up to week 52
  Anti-myotubularin TAb will be recorded from serum samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Gene Therapies
Locations (2):
- United States (2):
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.